CLINICAL TRIAL: NCT04480658
Title: Effectiveness of Bryophyllum Pinnatum by Patients With Nocturia and Its Effect on Sleep Quality
Brief Title: Effectiveness of Bryophyllum in Nocturia-Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01964
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Nocturia; Sleep Disorder
MeSH Terms: conditions — Nocturia; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bryophyllum pinnatum (Experimental): Bryophyllum pinnatum (BP) muscle relaxing substance
  Interventions: Drug: Bryophyllum pinnatum 50 %, tablets into capsules (verum: 2x2capsules/day)

INTERVENTIONS:
Drug: Bryophyllum pinnatum 50 %, tablets into capsules (verum: 2x2capsules/day) — Bryophyllum is administered for 3 weeks. Bryophyllum is given in form of capsules, 350mg per capsule, 0-0-2-2/d: 2 capsules 30min. before supper,2 capsules before going to bed.
  Other Names:
  Bryophyllum pinnatum/Kalanchoe

SUMMARY:
Night-time micturition, called nocturia, is a very common problem that unfavourably influences sleep- and life-qualities. The International Continence Society (ICS) defines nocturia as micturition once or several times during the night. Nocturia is one of the cardinal symptoms of overactive bladder (OAB). Persons with nocturia have the intention to continue sleep after going to the toilet which does not succeed to the same extent, depending on age.

The natural occurrence of the plant, Bryophyllum pinnatum (BP) which is used in this observational study origins from Madagascar as well as in tropical Africa, South America and Asia. In the folk medicine of these countries BP is widely used. BP has a calming, spasmolytic, anti-inflammatory, pain-relieving, diuretic and cytotoxic effects.

According to previous preclinical and clinical studies the inhibiting effect of BP on overactive bladder was proven. The pharmacological effect of this plant on uterine smooth muscle cells, on spontaneous and oxytocin-stimulated contractions, and on detrusor muscle cells in an in-vitro model of the pig's bladder was shown. Smooth muscle relaxation is not only required for preventing premature labour but also for symptom's relief of overactive bladder (OAB). The flavonoid, aglycons and bufadienolides, are components of the pressed juice of the BP leaves that have comparable effects to the standard drug oxybutynin on vesical smooth muscle cells.

Since many year BP is used in obstetrics not only as tocolytics but also as a sedative and sleeping pill.

There are known only few adverse events, such as skin irritation by intravenous application.

The interest in phytotherapeutical drugs for treatment the chronic diseases is very high and Bryophyllum is also frequently used in Switzerland for hyperactive conditions.

In Switzerland, following the vote on complementary medicine on 17.05.2009, alternative treatments will be covered by basic health insurance. Definitive inclusion in the catalogue of benefits will be granted if effectiveness, safety and cost-effectiveness can be demonstrated.

The potential and side-effect profile of BP, as well as the social interest in research into alternative methods is the background to the implementation of this observational study.

DETAILED DESCRIPTION:
In the therapeutic concept of the treatment of OAB, antimuscarinic drugs play a central role. Antimuscarinics are known to inhibit the contraction of detrusor muscle (smooth muscle cells) and block the muscarinic receptor (M2/M3) important for efferent nerve conduction. This conventional therapy for OAB can have important adverse effects, notably on the gastrointestinal tract with constipation, on the excretory glands in the sense of xerostomia/xerophthalmia, on the nerve cells of the brain inhibiting cognitive function and in the heart muscle cells accelerating the heart rate. Especially elderly people are affected by these undesirable effects. Because of changes in the receptor profile, the effect of antimuscarinics and improvement of symptoms might be lowered in elderly people and another substance with less side effects would be of great interest. No such adverse effects are reported for B. pinnatum. Until now, there are few data for its use in OAB. Efficacy and tolerability of B. pinnatum in the treatment of OAB are the major outcome measures of this clinical trial.

* 50 women are included in this observational study, treated with Bryophyllum pinnatum in form of the commercially available Bryophyllum tablets into capsules (verum: 2x2capsules/day). Recruitment time is planned from January, 2018 to January 2022.
* Duration of the drug administration is 3 weeks.
* Primary endpoint are the reduction of nocturia (measured by filling in a voiding dairy) and the change of sleep-quality (measured by using Pittsburgh Sleep Quality Index)
* secondary endpoints are the improvement of quality of life (measured by using the King's Health Questionnaire and the International Consultation on Incontinence Overactive Bladder Questionnaire (ICIQ-OAB), two questionnaires, validated for the German language and for women with incontinence), increase of the micturition volumes and reduction of urge episodes (measured by the patients and recorded in a voiding dairy) and the registration of adverse events during the study phase. Ethics committee approval has been given.

ELIGIBILITY:
Inclusion Criteria:

* Nocturia ≥2 Mal per a night
* Overactive bladder (>8 Mictions/day)
* Age > 18 Years
* local or systemic Therapy with Estrogen, if the therapy dates >4 Weeks before study-start.
* prior incontinence operation (if the operation dates back more than 6 months)
* german speaking Patients and a given informed consent

Exclusion Criteria:

* Intolerance against a substance or a compound
* participation in an other study 4 weeks prior to inclusion
* urinary tract infection
* drug abuse
* bladder affecting drugs like anticholinergics, diuretics, muscle relaxing medicaments and phytotherapeutics
* lactose intolerance
* Pregnant and lactating women
* Incompliance of Patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Reduction of nocturia frequency | 4 Weeks
  micturition protocol will be handed over during the baseline visit, it will be filled three days before the second visit in 1 week( therapy-start), follow-up control 3 weeks after medication intake and after the completed medication period ]
Sleep-Quality. | 4 Weeks
  Pittsburgh Sleep Quality Index (PSQI; score 0-21) will be handed over during the baseline visit and will be filled three days before the second visit in 1 Week and three days after the therapy-end (after 3 Weeks). The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

SECONDARY OUTCOMES:
Changes of overactive bladder symptoms | before the second visit in 1 week, at follow-up control 3 weeks after begin of medication intake and 4 weeks after end of medication intake.
  quality of life is measured by the ICIQ-OAB (score 0-16), a specific questionnaire for OAB
Safety of Bryophyllum: adverse events | 4 weeks
  during medication intake at 1 week and 3 weeks after start of medication intake, measured by a personal adverse event protocol
Daytime sleepiness | before the second visit in 1 week, at follow-up control 3 weeks after begin of medication intake and 4 weeks after end of medication intake.
  quality of life is measured by Epworth Sleepiness Scale Questionnaire (score 0-24)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hospital, Clinic for Gynecology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR